CLINICAL TRIAL: NCT04584242
Title: Prospective, Multicenter, Randomized, and Comparative Clinical Trials to Compare the Effects of Pioglitazone and Evogliptin on Hepatic Fibrosis in Patients With Chronic Hepatitis B With Significant Hepatic Fibrosis With Type 2 Diabetes
Brief Title: Clinical Trials to Compare the Effects of Pioglitazone and Evogliptin on Hepatic Fibrosis in Patients With Chronic Hepatitis B With Significant Hepatic Fibrosis With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0305
Record Dates: First submitted 2020-09-24; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Chronic Hepatitis B With Significant Hepatic Fibrosis With Type 2 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: gluconon tab 15mg
- Evogliptin (Experimental)
  Interventions: Drug: suganon tab 5mg

INTERVENTIONS:
Drug: gluconon tab 15mg — frosting and formulation : a round, convex tablet of white to gray. path of administration : once a day, two tabs, oral Amount of raw material medication (1 pill) : Pioglitazone hydrochloride 16.53mg storage method : Store 15 to 30°C to avoid light-tight containers and moisture manufacturing source : DONG-A ST
  Arms: Pioglitazone
Drug: suganon tab 5mg — frosting and formulation : pink circular film coating tablets path of administration : once a day, one tabs, oral Amount of raw material medication (1 pill) : Evogliptin tartrate 6.869mg(5mg as evogliptin) storage method : Confidential containers, stored at room temperature (1-30°C) manufacturing source : DONG-A ST
  Arms: Evogliptin

SUMMARY:
The clinical study determines the effect of Evogliptin in patients with type 2 diabetes mellitus and chronic hepatitis B to confirm the improvement of hepatic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Adultes between 20 and 80 years of age
* Patients who satisfy the following conditions among chronic hepatitis B patients diagnosed with type 2 diabetes

  1. Patients who are newly diagnosed as type 2 diabetes : 6.5% ≤ HbA1c < 10.0%
  2. Patients who are already diagnosed as type 2 diabetes: HbA1c < 10.0%
* Patients who have significant liver fibrosis of at least 7 kPa in a hepaticity test using fibroscan
* Patients who voluntarily signed the consent form after informed on the object, method, benefits and risks of the clinical study

Exclusion Criteria:

* Patients who were taking Pioglitazone or Evoglipitin medication or who took diabetes medication within 4 weeks at the time
* Patients who meet the standard of alcoholic fatty liver (in excess of 210g per week for men and 140g per week for women over the last two years)
* Liver cirrhosis patients with impaired liver function (CTP class B and C)
* Patients who took drugs that can cause fatty liver (amiodarone, methotrexate, tamoxifen, valproate, corticosteroids, etc.)
* Patients with acute or chronic metabolic acidosis with or without coma and history of ketonic acid (within 24 weeks)
* Allergic or hypersensitive to the target drug or its composition;
* Patients treated with oral or non - oral corticosteroid treatment for chronic (more than 14 consecutive days) within 8 weeks prior to screening.
* Poor nutrition, starvation, and debilitating conditions (including severe infections and severe injury patients before and after surgery)
* Patients who are receiving radiation and chemotherapy for malignant tumors or patients who have been on chemotherapy or radiation treatment for less than two years.
* Patients with heart failure in 24 weeks (class III to IV in NYHA classification) or unregulated arrhythmia.
* Patients with acute cardiovascular disease in 12 weeks or less (e.g. unstable angina, myocardial infarction, routine ischemic seizures, cerebrovascular disease, coronary bypass surgery, or coronary artery interventions).
* Patients with renal failure, chronic neuropathy (estimated glomerular filtration rate <60 mL/min/1.73 m2) or dialysis
* Anemia patients whose Hb levels are less than 10.5g/dl
* Women who are pregnant or breastfeeding
* Patients who do not agree to use proper contraception during clinical trials only for women or men.
* Patients who took medicines for clinical trials in other clinical trials within four weeks of document consent
* Patients who are unable to participate in clinical trials on the judgment of other researchers
* Patients who cannot read the consent form (e.g. illiteracy, foreigners, etc.)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline LSM (Liver Stiffness measurement) at week 24 (±7days) | Baseline
  Changes in the Liver Stiffness measurement after 24 weeks (±7days) compared to Baseline within and between arms
Changes from baseline LSM (Liver Stiffness measurement) at week 24 (±7days) | Baseline to 24 weeks (±7days)
  Changes in the Liver Stiffness measurement after 24 weeks (±7days) compared to Baseline within and between arms

SECONDARY OUTCOMES:
Changes from baseline CAP (Controlled Attenuation Parameter) at week 24 (±7days) within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Change from baseline at Week 24 (±7days) is defined as [(Baseline CAP value) - (Follow-up CAP value)] / (Baseline CAP value) * 100 (%)
Changes from baseline HbA1c at week 24 (±7days) within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Change from baseline at Week 24 (±7days) is defined as HbA1c at Week 24 (±7days) minus HbA1c at Week 0
Changes from baseline Insulin at week 24 (±7days) within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Change from baseline at Week 24 (±7days) is defined as insulin at Week 24 (±7days) minus insulin at Week 0
Changes from baseline lipid profile (total cholesterol, HDL, LDL, TG) at week 24 (±7days) within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Change from baseline at Week 24 (±7days) is defined as lipid profile (total cholesterol, HDL, LDL, TG) at Week 24 (±7days) minus lipid profile at Week 0
Changes from baseline AST/ALT at week 24 (±7days) within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Change form baseline at Week 24 (±7days) is defined as the proportion of AST/ALT values who are normalized at Week 24 (±7days)
Changes from baseline Body weight at week 24 (±7days) within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Change from baseline at Week 24 (±7days) is defined as body weight at Week 24 minus body weight at Week 0
Changes from baseline Liver fibrosis and fatty liver at week 24 (±7days) among the MRE+MRI PDFF enforcement arms within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Change from baseline at Week 24 (±7days) is defined by MRE+MRI PDFF
Proportions of adverse effects and drug interruptions or changes between baseline and week 24 (±7days) within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Compare between baseline at Week 24 (±7days) is defined as the occurrence rate of adverse events and drug interruptions or changes
Prognostic factor of the Improvement of Liver fibrosis between baseline and week 24 (±7days) within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Prediction Factor Analysis of the Improvement of Liver fibrosis after 24 (±7days) weeks compared to Baseline within and between arms
Prognostic factor of the Improvement of Fatty liver between baseline and week 24 (±7days) within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Prediction Factor Analysis of the Improvement of Fatty liver after 24 weeks (±7days) compared to Baseline within and between arms
Prognostic factor of the Improvement of HbA1 between baseline and week 24 (±7days) within and between arms | 1) Baseline, 2) Baseline to 24 weeks (±7days)
  Prediction Factor Analysis of the Improvement of HbA1c after 24 weeks (±7days) compared to Baseline within and between arms

CONTACTS AND LOCATIONS:
Overall Officials: Seung Up Kim, Principal Investigator — Severance Hospital
Locations (4):
- South Korea (4):
  - Gangnam Severance Hospital, Seoul
  - Samsung Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No